CLINICAL TRIAL: NCT03106896
Title: Involvement of Reorganization of Cerebral Functional Connectivity in the Process of Transition to Postherpetic Neuralgia
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Sponsor
Other Study IDs: 2016-069
Record Dates: First submitted 2017-03-26; First posted 2017-04-11 (Actual); Last update posted 2017-04-11 (Actual); Status verified 2016-12

CONDITIONS: Postherpetic Neuralgia
MeSH Terms: conditions — Neuralgia, Postherpetic

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

GROUPS / COHORTS (3):
- postherpetic neuralgia (PHN group): persist more than 3 months after the resolution of the acute shingles episode and have pain intensity greater than 4 on the visual analog scale (VAS 0, no pain; 10, "worst pain imaginable").
- acute herpetic pain (AHP group): have pain (VAS≧4 ) duration of within 7 days after zoster onset at initial interview
- healthy control (CON group): healthy population

SUMMARY:
Postherpetic neuralgia(PHN) is a chronic neuropathic pain syndrome which persists more than 3 months after the resolution of the acute shingles episode. PHN is a complicated neuropathic pain that results from the sustained peripheral injury by herpes zoster and its pathological mechanism in skin and spine has been reported. But the cerebral mechanism is still unclear. Based on the previous study that has proved the reorganization of cerebral functional connectivity in pain chronicity, the investigators hypothesize that the process from acute herpetic pain (AHP) to PHN is also accompanied with the reorganization of functional connectivity.In the study, the investigators intend to use 7 Tesla functional magnetic resonance imaging(fMRI) to observe the difference of brain activity and functional connectivity between acute herpetic pain and PHN. Meanwhile, the investigators examine the evolution of functional connectivity longitudinally in patients who is suffering from acute pain, so as to explore the central mechanism of transition to PHN.

DETAILED DESCRIPTION:
Postherpetic neuralgia(PHN) is a chronic neuropathic pain syndrome which persists more than 3 months after the resolution of the acute shingles episode. PHN is the most common complication of herpes zoster in the pain clinic and it was reported that 2%-35% patients who suffer from herpes zoster may continue to suffer from PHN. Along with the coming of aging population, advanced age is one of the risk factors and about 20.6% patients aged 50 years and over may translate into PHN from acute herpes zoster . Besides, the proportion may increase with age which not only seriously impacts the quality of patients' life but also causes huge personal and social healthcare burden.

PHN is a complicated neuropathic pain that results from the sustained peripheral injury by herpes zoster and its pathological mechanism in skin and spine has been reported. But the cerebral mechanism is still unclear. In the recent several years, fMRI is widely used in the cerebral mechanism in several diseases due to its no trauma and accurate positioning about brain regions. The existing fMRI research about PHN discovered that the alteration of brain activity and reorganization of cerebral functional connectivity in PHN compared with healthy subjects. Liu,et al. investigated the effects of PHN on resting-state brain activity utilizing arterial spin labeling (ASL) techniques and found that regional cerebral blood flow in left caudate, left insula, left S1, and right thalamus was highly correlated with the pain intensity, and meanwhile, the four brain regions exist functional connectivity with other regions in different degrees. Liang,et al. explored the difference of cerebral activity between acute herpes zoster and PHN and found PHN showed higher regional homogeneity in bilateral thalamus, right cerebellum, right hippocampus, right fusiform gyrus, right insula. They speculated tha the thalamus, cerebellum, insula may be associated with hyperalgesia and hippocampus may be associated with pain memory in PHN patients.

In conclusion, fMRI showed that insula, thalamus, hippocampus, striatum and so on are connected with PHN. And then the investigators are curious about the cerebral alteration before the patient is definitely diagnosed as PHN. Meanwhile it's commonly presented in clinic that why some patients who suffer from herpes zoster can heal without PHN while someone are suffering from PHN in a long time. The investigators assume that cerebral alteration and its functional connectivity are associated with the transition to PHN. That is to say, it's a study of mechanism about the transition from acute herpes zoster pain to PHN. Some studies have shown that the reorganization of neural network, especially the function connectivity between cortex and limbic system, is involved in the transition to chronic back pain and affects the sense, emotion, cognition, movement of pain. Apkarian ,et al. used fMRI to identify intrinsic and extrinsic hippocampal functional connectivity, comparing subacute back pain (SBP, back pain 1-4 mo) and chronic back pain (CBP, back pain﹥1 yr) patients to control subjects. Both groups showed more extensive hippocampal connectivity than CON subjects. They then examined the evolution of hippocampal connectivity longitudinally in SBP patients who recovered (SBPr, back pain decreased﹥20% in 1 yr) and those with persistent pain (SBPp) and found that SBPp and SBPr subjects have distinct changes in hippocampal-cortical connectivity over 1 yr. Specifically, SBPp subjects showed large decreases in hippocampal connectivity with medial prefrontal cortex. These results demonstrated that the reorganization of hippocampal functional connectivity is associated with the transition to chronic back pain. They also found that nucleus accumbens(NAc)-medial prefrontal cortex(mPFC) functional connectivity is also involved in the transition to chronic back pain.

So the investigators hypothesize that the process from acute herpetic pain (AHP) to PHN is also accompanied with the reorganization of functional connectivity.

With the development of technology, 7 Tesla fMRI is coming into our sight. Andreas, et al. showed that 7 Tesla-fMRI with the increased field strength offers marked improvement for the localization of activation foci with high spatial specificity when comparing neural response to painful electrical stimulation with 3 Tesla. In our study, the investigators intend to use 7 Tesla fMRI to observe the difference of brain activity and functional connectivity between acute herpetic pain and PHN. Meanwhile, the investigators examine the evolution of functional connectivity longitudinally in patients who is suffering from acute pain, so as to explore the central mechanism of transition to PHN.

ELIGIBILITY:
Inclusion Criteria:

* All participants are more than 50 years old, right-handed. Patients are definitely diagnosed by a clinician for postherpetic neuralgia (PHN), persisting pain more than 3 months after the resolution of the acute shingles episode and have pain intensity greater than 4 on the visual analog scale (VAS 0, no pain; 10, "worst pain imaginable"). Patients who are diagnosed as acute herpes zoster at the initial interview have pain (VAS≧4 ) duration of within 7 days after zoster onset. Data are available for healthy control subjects with age and sex matched.

Exclusion Criteria:

* Subjects are excluded if they are suffering from eyes, ears, viscera, meninx herpes zoster and asymptomatic special herpes zoster. Those who report any other acute and chronic painful conditions, systemic disease, history of head injury, psychiatric diseases, or more than mild depression [(score > 19, according to Beck's Depression Inventory (BDI)] are also excluded. Subjects are excluded if they were found abnormal signal when scanning by fMRI and exist MRI contraindication, such as existence of magnetic metal in body, claustrophobia and so on. Patients who don't withdraw the analgesic medication (oxycodone, NSAIDS, gabapentin, etc.) the day before and on the day of examination are also excluded.

Ages: 50 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The PHN sample size is determined according to the published reports. The AHP sample size is determined according to the 20.6% incidence of patients who translate from AHP to PHN and the drop-out rate, generally speaking, about 10%. Finally, we determine we need 54 AHP subjects, 10 PHN subjects, 11 age and gender-matched control subjects.
Sampling Method: Probability Sample
Enrollment: 75 (Estimated)
Dates: Start 2017-04 (Estimated); Primary Completion 2020-06 (Estimated); Study Completion 2020-06 (Estimated)

PRIMARY OUTCOMES:
functional connectivity between several brain regions | AHPand CON subjects are scanned at four visits over the course of six months to observe the variation trend of connectivity from the AHP to PHN. PHN group need only one scanning.
  The functional connectivity between several brain regions in AHP group and PHN group is different. Besides, the reorganization of cerebral functional connectivity in the process of transition to postherpetic neuralgia is relevant with the chronicity of symptom.

IPD SHARING:
Plan to Share IPD: No